CLINICAL TRIAL: NCT06587997
Title: Changes in Renal Perfusion During Hemodialysis in Patients with End-stage Renal Disease: a Prospective Observational Study
Brief Title: Changes in Renal Perfusion During Hemodialysis in Patients with End-stage Renal Disease
Acronym: HD-RPC
Status: Not yet recruiting | Type: Observational
Sponsor: Yuanjun Yang (Other)
Responsible Party: Sponsor-Investigator, Yuanjun Yang, Director, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: HD-RPC
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: End-stage Renal Disease
Keywords: hemodialysis; renal perfusion; end-stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Residual renal function (RRF) characteristically declines after patients with end-stage renal disease (ESRD) initiate dialysis. Although RRF preservation correlates with improved patient's quality of life and survival prospects, poor understanding of the pathophysiology underlying RRF decline limits protection strategies.

DETAILED DESCRIPTION:
Hemodialysis (HD) is the primary renal replacement therapy for patients with end-stage renal disease. However, residual renal function (RRF) characteristically declines after these individuals start dialysis. This loss of RRF not only impacts the adequacy of dialysis and control of complications but also affects the patient's quality of life and survival prospects. Due to a lack of clear understanding regarding the pathophysiology underlying this decline in RRF, no effective strategies exist for its preservation at present. The objective of this study is to explore the changes in renal perfusion during hemodialysis in patients with end-stage renal disease, and provide a new idea for protection of RRF. This study was an observational study, and no interventions were performed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Clinical diagnosis of end-stage renal disease requiring long-term hemodialysis treatment, with dialysis duration ≤ 3 months;
* Urine output > 500ml/day or GFR > 3ml/min/1.72m2;
* Signed and dated informed consented is obtained.

Exclusion Criteria:

* Presence of vascular access dysfunction (blood flow rate < 180ml/min);
* Severe heart failure;
* Active infection;
* Infectious disease;
* Patients with severe anemia;
* Patients with polycystic kidney disease;
* Expected dialysis duration < 6 months;
* Pregnancy or lactation women;
* Patients who are participating in other clinical studies, or who have participated in other clinical studies within 3 months prior to enrollment;
* Unwillingness to be followed up or poor adherence to treatment;
* Other circumstances that the investigator considers unsuitable for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First Medical Center of Chinese PLA General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-09-05 (Estimated); Primary Completion 2026-09-03 (Estimated); Study Completion 2026-09-03 (Estimated)

PRIMARY OUTCOMES:
renal perfusion | one day
  Changes in renal perfusion during hemodialysis in patients with end-stage renal disease

SECONDARY OUTCOMES:
diastolic blood pressure | one day
  diastolic blood pressure during hemodialysis in patients with end-stage renal disease
systolic blood pressure | one day
  systolic blood pressure during hemodialysis in patients with end-stage renal disease
urine volume | 10 months
  Urine volume within 10 months of starting dialysis